CLINICAL TRIAL: NCT00413179
Title: The Effect of Metformin Added to Clomiphene Citrate on Pregnancy Rates in Hyperandrogenic, Chronic Oligoovulatory or Anovulatory Women: A Randomized Trial
Brief Title: The Effect of Metformin Added to Clomiphene Citrate on Pregnancy Rates in Hyperandrogenic, Chronic Oligoovulatory or Anovulatory Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWH19970383H
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2006-12-19 (Estimated); Status verified 2006-12

CONDITIONS: Polycystic Ovary Syndrome; Anovulation; Oligoovulation; Infertility; Hyperandrogenism
Keywords: Polycystic Ovarian Syndrome; Chronic Anovulation; Chronic Oligoovulation; Infertility; Hyperandrogenism; Metformin; Ovulation induction
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation; Infertility; Hyperandrogenism | interventions — Metformin; Clomiphene

INTERVENTIONS:
Drug: Metformin
Drug: Clomiphene citrate
Drug: Placebo

SUMMARY:
The purpose of our study was to conduct a placebo controlled, double-blind randomized trial in chronic oligoovulatory or anovulatory , hyperandrogenic, infertility patients comparing the effects of adjuvant metformin plus clomiphene citrate to clomiphene citrate plus placebo on pregnancy rates and ovulation rates. We hypothesized that combining metformin with clomiphene citrate would result in higher ovulation and pregnancy rates in hyperandrogenic women who have chronic oligoovulation or anovulation as the sole etiology for their infertility and who have unknown responsiveness to clomiphene citrate.

DETAILED DESCRIPTION:
Women with polycystic ovary syndrome (PCOS), defined as chronic oligoovulation or anovulation and hyperandrogenism, are primarily treated with clomiphene citrate as first line therapy if they desire pregnancy. However, women with PCOS have lower than expected pregnancy rates in response to clomiphene citrate. Approximately 20% of women with PCOS are resistant to clomiphene citrate. Subjects with chronic oligoovulation or anovulation and hyperandrogenism will ovulate 80% of the time, but pregnancy occurs in only 40%. The ideal initial treatment regimen for women with PCOS who desire pregnancy has not been determined.

Metformin (Glucophage; Bristol-Myers Squibb, Princeton, NJ) is an insulin sensitizer and lowers serum insulin and androgen levels. Numerous case studies, case series, retrospective studies, and non-placebo controlled prospective studies, have suggested an improvement in insulin sensitivity, spontaneous menses, ovulatory response and pregnancies when metformin was given alone or prior to initiation of ovulation inducing agents in women with chronic anovulation and hyperandrogenism.

However, there has been conflicting evidence in the literature regarding the effect of metformin alone or in combination with ovulation inducing agents regarding ovulation and pregnancy rates in prospective, randomized trials. Therefore, it remains unknown if the use of metformin plus clomiphene citrate in non-selected, infertility patients with PCOS improves ovulation and pregnancy rates compared to the use of clomiphene citrate alone.

Women with a history of infertility and diagnosed with hyperandrogenic, oligoovulatory or anovulatory cycles as the sole etiology for their infertility were randomized to receive clomiphene citrate 50 mg days 5-9, plus metformin 500 mg three times daily versus clomiphene plus placebo. The dose of clomiphene was increased up to a maximum dose of 250 mg in a step-wise fashion until ovulation was confirmed with an ovulation predictor kit. Once ovulation was confirmed the subjects continued the ovulatory dose of clomiphene for 6 ovulatory cycles or until conception. Metformin or placebo was started on cycle day one and discontinued 8 days after the LH surge and/or by cycle day 21. A positive HCG, ovulation rates and pregnancy outcome were the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Married
* Hyperandrogenic women 18-40 years old who desired fertility and who demonstrated chronic anovulation or oligoovulation
* Had patent fallopian tubes and whose partners had normal semen analyses were eligible for enrollment in the study.

Exclusion Criteria:

* Androgen secreting tumours
* Diabetes mellitus
* Thyroid abnormalities
* Hyperprolactinemia
* Adult onset congenital adrenal hyperplasia
* Diminished ovarian reserve
* Subjects who used hormonal medications two months prior to the start of the trial.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56
Dates: Start 1997-12; Study Completion 2003-04

PRIMARY OUTCOMES:
Pregnancy Rates
Ovulation Rates

SECONDARY OUTCOMES:
Pregnancy Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Randal D Robinson, MD, Principal Investigator — Wilford Hall Medical Center and Brooke Army Medical Center
Locations (1):
- Wiford Hall Medical Center, Lackland Air Force Base, Texas, United States